CLINICAL TRIAL: NCT01666470
Title: Quality of Life of Patients With a History of Drug Allergy in Thailand
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Jettanong Klaewsongkram, Head of Division of Allergy and Clinical Immunology, Department of Medicine, Chulalongkorn University
Other Study IDs: Chula-ARC 001/12
Record Dates: First submitted 2012-08-12; First posted 2012-08-16 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Quality of Life
Keywords: Quality of life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug allergy patients: Patients with a history of drug allergy in Thailand
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — DrHy-Q (Thai version) and WHOQOL-BREF-THAI will be asked

SUMMARY:
Quality of life of patients with a history of drug allergy in Thailand will be studied.

DETAILED DESCRIPTION:
Thai patients with a history of drug allergy will be evaluated for their quality of life based on drug hypersensitivity quality of life questionnaire (DrHy-Q; Thai version) and The World Health Organization Quality of Life instrument (WHOQOL-BREF-THAI)

ELIGIBILITY:
Inclusion Criteria:

* Have a history of drug allergy
* At least 18 years of age

Exclusion Criteria:

* Not be able to understand Thai language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patients with a history of drug allergy
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The quality of life of Thai patients with a history of drug allergy evaluating by DrHy-Q (Thai version) | 1 year

SECONDARY OUTCOMES:
The correlation between DrHy-Q (Thai version) and WHOQOL-BREF-THAI | 1 year
  Pearson correlation coefficient between scores from DrHy-Q (Thai version) and WHOQOL-BREF-THAI in patients with a history of drug allergy will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Chulalongkorn University, Bangkok
  - Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok

REFERENCES:
- See also: Reliability and validity of the Thai Drug Hypersensitivity Quality of Life Questionnaire: a multi-center study — https://www.ncbi.nlm.nih.gov/pubmed/30346532